CLINICAL TRIAL: NCT04072315
Title: A Phase 2a Evaluation of PLN-74809 on αvβ6 Receptor Occupancy Using PET Imaging in Participants With IPF
Brief Title: Phase 2a Evaluation of PLN-74809 on αvβ6 Receptor Occupancy Using PET Imaging in Participants With IPF/
Acronym: IPF-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pliant Therapeutics, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PLN-74809-IPF-201
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Open label, incomplete crossover, up to 2 single doses administered at two different times
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PLN-74809 Dose Level 1 (60 mg) (Experimental): PLN-74809 Dose Level 1 (60mg)
  Interventions: Drug: PLN-74809; Radiation: Knottin tracer
- PLN-74809 Dose Level 2 (80 mg) (Experimental): PLN-74809 Dose Level 2 (80 mg)
  Interventions: Drug: PLN-74809; Radiation: Knottin tracer
- PLN-74809 Dose Level 3 (120 mg) (Experimental): PLN-74809 Dose Level 3 (120 mg)
  Interventions: Drug: PLN-74809; Radiation: Knottin tracer
- PLN-74809 Dose Level 4 (240 mg) (Experimental): PLN-74809 Dose Level 4 (240 mg)
  Interventions: Drug: PLN-74809; Radiation: Knottin tracer
- PLN-74809 Dose Level 4 (320 mg) (Experimental): PLN-74809 Dose Level 4 (320 mg)
  Interventions: Drug: PLN-74809; Radiation: Knottin tracer

INTERVENTIONS:
Drug: PLN-74809 — PLN-74809
Radiation: Knottin tracer — Radiotracer

SUMMARY:
A study in mild/moderate IPF patients using an αVβ6 PET ligand to evaluate target engagement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF, within 5 years prior to Screening,
* FVC %predicted ≥45%; historical FVC for entry in the study is permitted if within 1 month of screening.
* DLco (hemoglobin-adjusted) ≥30%; historical DLco for entry in the study is permitted if within 1 month of screening.
* Participants receiving treatment for IPF with nintedanib or pirfenidone are allowed,if on a stable dose for at least 3 months

Exclusion Criteria:

* Currently receiving or planning to initiate treatment for IPF (fibrosis) with agents not approved for that indication by the FDA
* Forced expiratory volume during the first seconds of the forced breath (FEV1)/FVC ratio <0.7
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis that can affect FVC measurement or IPF progression
* Known acute IPF exacerbation or suspicion by the Investigator of such, within 6 months of Screening
* Smoking of any kind within 3 months of Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics Medical Monitor, Study Director — Pliant Therapeutics, Inc.
Locations (1):
- Stanford Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mooney JJ, Jacobs S, Lefebvre EA, Cosgrove GP, Clark A, Turner SM, Decaris M, Barnes CN, Jurek M, Williams B, Duan H, Kimura R, Rizzo G, Searle G, Wardak M, Guo HH. Bexotegrast Shows Dose-Dependent Integrin alphavbeta6 Receptor Occupancy in Lungs of Participants with Idiopathic Pulmonary Fibrosis: A Phase 2, Open-Label Clinical Trial. Ann Am Thorac Soc. 2025 Mar;22(3):350-358. doi: 10.1513/AnnalsATS.202409-969OC. PMID 39499805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant on this study was enrolled in February 2020 and the last participant in May 2022. The enrollment period was prolonged due to the limited clinical trial operations at the research site, caused by COVID-19 pandemic.
Groups:
- 60 mg: PLN-74809: PLN-74809 (60 mg)
  Knottin tracer: Radiotracer
- 120 mg and 240 mg: PLN-74809: PLN-74809 (120 mg and 240 mg)
  Knottin tracer: Radiotracer
- 320 mg: PLN-74809: PLN-74809 (320 mg)
  Knottin tracer: Radiotracer
- 240 mg and 320 mg: PLN-74809: PLN-74809 (240 mg and 320 mg)
  Knottin tracer: Radiotracer
- 320 mg and 120 mg: PLN-74809: PLN-74809 (320 mg and 120 mg)
  Knottin tracer: Radiotracer
- 80 mg and 240 mg: PLN-74809: PLN-74809 (80 mg and 240 mg)
- 80 mg and 120 mg: PLN-74809: PLN-74809 (80 mg and 120 mg)
- 120 mg and 320 mg: PLN-74809: PLN-74809 (120 mg and 320 mg)
Period: Overall Study
Arm/Group | 60 mg | 120 mg and 240 mg | 320 mg | 240 mg and 320 mg | 320 mg and 120 mg | 80 mg and 240 mg | 80 mg and 120 mg | 120 mg and 320 mg
Started | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 60 mg: PLN-74809: PLN-74809 (60 mg)
- 120 mg and 240 mg: PLN-74809: PLN-74809 (120 mg and 240 mg)
- 320 mg: PLN-74809: PLN-74809 (320 mg)
- 240 mg and 320 mg: PLN-74809: PLN-74809 (240 mg and 320 mg)
- 320 mg and 120 mg: PLN-74809: PLN-74809 (320 mg and120 mg)
- Total: Total of all reporting groups
Arm/Group | 60 mg | 120 mg and 240 mg | 320 mg | 240 mg and 320 mg | 320 mg and 120 mg | 80 mg and 240 mg | 80 mg and 120 mg | 120 mg and 320 mg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77 (0) | 69 (0) | 76 (0) | 83.5 (.71) | 77 (0) | 76 (0) | 77 (0) | 79 (0) | 77.6 (4.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Male | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Predicted Effect on αVβ6 PET ( Positron Emission Tomography) in Lungs After Administration of Drug.
Description: Assessment of the primary endpoint was made using standard methods for quantifying the amount to PET tracer bound to the αvβ6 integrin receptor in the lungs before and after administration of study drug and PK/PD modeling.
Time Frame: Following 1 day of dosing
Measure: Count of Participants; unit: Participants
Groups:
- 80 mg and 240 mg: PLN-74809: PLN-74809 (80 mg and 240 mg)
  Knottin tracer: Radiotracer
- 80 mg and 120 mg: PLN-74809: PLN-74809 (80 mg and 120 mg)
  Knottin tracer: Radiotracer
- 120 mg and 320 mg: PLN-74809: PLN-74809 (120 mg and 320 mg)
  Knottin tracer: Radiotracer
Arm/Group | 60 mg | 120 mg and 240 mg | 320 mg | 240 mg and 320 mg | 320 mg and 120 mg | 80 mg and 240 mg | 80 mg and 120 mg | 120 mg and 320 mg
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Participants | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1

2. Secondary Outcome: Safety and Tolerability of PLN-74809 as Measured by the Number / Percentage of Adverse Events
Description: Adverse events were collected from the time the participant signs the Informed Consent Form until the last day of visit (Day 14).
Time Frame: From screening to 1 week following the administration of PLN-74809
Measure: Count of Participants; unit: Participants
Groups:
- 320 mg and 120 mg: PLN-74809: PLN-74809 (320 mg and 120 mg)
Arm/Group | 60 mg | 120 mg and 240 mg | 320 mg | 240 mg and 320 mg | 320 mg and 120 mg | 80 mg and 240 mg | 80 mg and 120 mg | 120 mg and 320 mg
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 Days
Groups:
- 60 mg: PLN-74809 (60 mg)
- 120 mg and 240 mg: PLN-74809 (120 mg and 240 mg)
- 320 mg: PLN-74809 (320 mg)
- 240 mg and 320 mg: PLN-74809 (240 mg and 320 mg)
- 320 mg and 120 mg: PLN-74809 (320 mg and 120 mg)
- 80 mg and 240 mg: PLN-74809 (80 mg and 240 mg)
- 80 mg and 120 mg: PLN-74809 (80 mg and 120 mg)
- 120 mg and 320 mg: PLN-74809 (120 mg and 320 mg)
Arm/Group | 60 mg | 120 mg and 240 mg | 320 mg | 240 mg and 320 mg | 320 mg and 120 mg | 80 mg and 240 mg | 80 mg and 120 mg | 120 mg and 320 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 0/2 | 0/1 | 1/1 | 0/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg (N=1) | 120 mg and 240 mg (N=1) | 320 mg (N=1) | 240 mg and 320 mg (N=2) | 320 mg and 120 mg (N=1) | 80 mg and 240 mg (N=1) | 80 mg and 120 mg (N=1) | 120 mg and 320 mg (N=1)
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Elevated Gamma Glutamyl Transferase
Hepatic Enzyme Increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Elevated liver enzymes (AST, ALT, AlkP'tase)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT04072315/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT04072315/SAP_001.pdf